CLINICAL TRIAL: NCT03413878
Title: Snow Properties and Its Modeling for Studying Gas Exchange Under the Simulated Avalanche Snow
Acronym: SPAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Czech Technical University in Prague (Other)
Collaborators: Charles University, Czech Republic (Other); Ministry of Defence and Armed Forces of the Czech Republic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: VentRes-2018-01-KR
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Accident Caused by Snow Avalanche
Keywords: snow; avalanche; hypercapnia; work of breathing
MeSH Terms: conditions — Hypercapnia | interventions — Respiration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Wet snow/Small air pocket (Experimental): Breathing in the simulated avalanche snow. Breathing into model of wet avalanche snow with a small air pocket
  Interventions: Other: Breathing in the simulated avalanche snow
- Dry snow/Small air pocket (Experimental): Breathing in the simulated avalanche snow. Breathing into model of dry avalanche snow with a small air pocket
  Interventions: Other: Breathing in the simulated avalanche snow
- Wet snow/Large air pocket (Experimental): Breathing in the simulated avalanche snow. Breathing into model of wet avalanche snow with a large air pocket
  Interventions: Other: Breathing in the simulated avalanche snow
- Dry snow/Large air pocket (Experimental): Breathing in the simulated avalanche snow. Breathing into model of dry avalanche snow with a large air pocket
  Interventions: Other: Breathing in the simulated avalanche snow

INTERVENTIONS:
Other: Breathing in the simulated avalanche snow — Breathing in the simulated wet or dry avalanche snow with a small or large air pocket

SUMMARY:
The aim of the study is to investigate respiratory parameters of a person in the simulated avalanche snow and consequent use of the measured data for development of a mathematical-physical model of breathing during increasing hypercapnia in the avalanche.

DETAILED DESCRIPTION:
The study is a part of a university research project aimed at studying physiological conditions and development of breathing parameters of a person breathing in the simulated avalanche snow. Presence of an air pocket and its size play an important role in survival of victims buried in the avalanche snow. Even small air pockets facilitate breathing, yet they do not provide a significant amount of fresh air for breathing. The investigators hypothesize that the size of the air pocket significantly affects the airflow resistance and work of breathing. The aim of the study is to investigate the effect of the air pocket volume on gas exchange and work of breathing in subjects breathing into the simulated avalanche snow.

ELIGIBILITY:
Inclusion Criteria:

* healthy and fit volunteers, classified as The American Society of Anesthesiologists class I
* without a smoking history

Exclusion Criteria:

* Tiffeneau Index less than 0.70
* any cardiovascular or respiratory condition

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-01-29 (Actual); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-05-20 (Estimated)

PRIMARY OUTCOMES:
The length of breathing | Continuously within 30 minute interval from the beginning of the breathing experiment
  Time to termination of the breathing experiment due to the decision of the tested subject, or determined by high end-tidal carbon dioxide value or by the order by the clinician assessing the health status of the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubik, PhD, Principal Investigator — Czech Technical University in Prague, FBMI
Locations (2):
- Czechia (2):
  - Czech Technical University, Faculty of Biomedical Engineering, Kladno
  - Charles University, Czech Republic, Prague

REFERENCES:
- [Background] Brugger H, Sumann G, Meister R, Adler-Kastner L, Mair P, Gunga HC, Schobersberger W, Falk M. Hypoxia and hypercapnia during respiration into an artificial air pocket in snow: implications for avalanche survival. Resuscitation. 2003 Jul;58(1):81-8. doi: 10.1016/s0300-9572(03)00113-8. PMID 12867313
- [Background] Bellani G, Patroniti N, Weismann D, Galbiati L, Curto F, Foti G, Pesenti A. Measurement of pressure-time product during spontaneous assisted breathing by rapid interrupter technique. Anesthesiology. 2007 Mar;106(3):484-90. doi: 10.1097/00000542-200703000-00012. PMID 17325506
- [Background] Grissom CK, Radwin MI, Harmston CH, Hirshberg EL, Crowley TJ. Respiration during snow burial using an artificial air pocket. JAMA. 2000 May 3;283(17):2266-71. doi: 10.1001/jama.283.17.2266. PMID 10807386
- [Background] Roubik K, Sieger L, Sykora K. Work of Breathing into Snow in the Presence versus Absence of an Artificial Air Pocket Affects Hypoxia and Hypercapnia of a Victim Covered with Avalanche Snow: A Randomized Double Blind Crossover Study. PLoS One. 2015 Dec 14;10(12):e0144332. doi: 10.1371/journal.pone.0144332. eCollection 2015. PMID 26666523
- [Background] Strapazzon G, Paal P, Schweizer J, Falk M, Reuter B, Schenk K, Gatterer H, Grasegger K, Dal Cappello T, Malacrida S, Riess L, Brugger H. Effects of snow properties on humans breathing into an artificial air pocket - an experimental field study. Sci Rep. 2017 Dec 15;7(1):17675. doi: 10.1038/s41598-017-17960-4. PMID 29247235
- [Derived] Roubik K, Sykora K, Sieger L, Ort V, Horakova L, Walzel S. Perlite is a suitable model material for experiments investigating breathing in high density snow. Sci Rep. 2022 Feb 8;12(1):2070. doi: 10.1038/s41598-022-06015-y. PMID 35136116
- See also: Work of Breathing into Snow in the Presence versus Absence of an Artificial Air Pocket Affects Hypoxia and Hypercapnia of a Victim Covered with Avalanche Snow: A Randomized Double Blind Crossover Study — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0144332